CLINICAL TRIAL: NCT03615781
Title: Two Versus Four Weeks of Antibiotic Treatment in Native Joint Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilker Uckay, Attending, Docent Dr. med Ilker Uçkay, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: no. 15-014
Record Dates: First submitted 2017-01-16; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Arthritis, Septic
Keywords: septic arthritis; surgery; antibiotic duration; remission; sequelae
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Two week's arm - surgery (Experimental): The investigators perform a surgical drainage and removal of the infected orthopedic implant.
  Interventions: Procedure: Two week's arm - surgery
- Four week's arm - surgery (Active Comparator): The investigators surgically remove the infected implant.
  Interventions: Procedure: Four week's arm - surgery
- Two week's arm - drugs (Experimental): The investigators perform a surgical drainage and removal of the infected orthopedic implant. They start an empirical antibiotic treatment based on patient's history and co-morbidities, such as vancomycin or amoxicillin/clavulanic acid. The adapt later on the targeted antibiotic therapy according to the causative pathogens and their antibiotic susceptibility testing.
  Interventions: Drug: Two week's arm - drugs
- Four week's arm - drugs (Active Comparator): The investigators surgically remove the infected implant and all soft tissue infection. Instead of a total of 2 week's of antibiotic therapy, they administer a total of 4 weeks of systemic antibiotic therapy targeted to the pathogen(s).
  Interventions: Drug: Four week's arm - drugs

INTERVENTIONS:
Procedure: Two week's arm - surgery — The investigators perform a surgical drainage of the infection along with the complete removal of the infected orthopedic implant.
  Arms: Two week's arm - surgery
Procedure: Four week's arm - surgery — The investigators perform a surgical drainage of the infection along with the complete removal of the infected orthopedic implant.
  Arms: Four week's arm - surgery
Drug: Two week's arm - drugs — After the surgical implant removal, the investigators prescribe a total of 2 weeks of systemic targeted antibiotic therapy against the causative pathogen(s), of which one week is recommended to be intravenously.
  Arms: Two week's arm - drugs
Drug: Four week's arm - drugs — After the surgical implant removal, the investigators prescribe a total of 4 weeks of systemic targeted antibiotic therapy against the causative pathogen(s), of which one week is recommended to be intravenously.
  Arms: Four week's arm - drugs

SUMMARY:
The optimal duration of systemic antibiotic administration for native joint septic arthritis is unknown. The investigators perform a randomized study allowing up to 3 surgical lavages and allocating patients into a two-week's and a four week's randomization arm

DETAILED DESCRIPTION:
The optimal duration of systemic antibiotic administration for native joint septic arthritis is unknown. The investigators perform a randomized study allocating patients into a two-week's and a four week's randomization arm.

The adult patients are hospitalized for septic arthritis. A computer program randomizes 1:1 between a two week's and a four week's arm of targeted antibiotic treatment of which at least the first week is intravenously. The randomization may occur until Day 5 of admission. Up to three surgical interventions are allowed. The investigators allow the inclusion of all bacterial arthritis and all joints.

ELIGIBILITY:
Inclusion Criteria:

1. Age >17 years
2. Microbiologically-confirmed septic arthritis
3. At least one surgical drainage/lavage

Exclusion Criteria:

1. Presence of osteosynthesis material in the vicinity of the articulation
2. Presence of a concomitant infection needing more than 2 week's of antibiotic therapy
3. More than 3 surgical drainages
4. Life expectancy less than 6 months
5. Chronic osteomyelitis in vicinity of the arthritis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical Remission of systemic infection | 6 months
  Measurement of fever.
Sequels | 6 months
  Patient's remaining gait disorders.
  * range of movement in adjacent joints of former infection
  * questionnaire regarding persistant pain and handicaps (open wording)

SECONDARY OUTCOMES:
Wound redness | 6 months
  Visual examination of the presence of wound redness.
Wound discharge | 6 months
  Visual examination of the presence of wound discharge
Presence of pus | 6 months
  Visual examination of the presence of pus coming out the wound

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uckay I, Tovmirzaeva L, Garbino J, Rohner P, Tahintzi P, Suva D, Assal M, Hoffmeyer P, Bernard L, Lew D. Short parenteral antibiotic treatment for adult septic arthritis after successful drainage. Int J Infect Dis. 2013 Mar;17(3):e199-205. doi: 10.1016/j.ijid.2011.12.019. Epub 2012 Nov 22. PMID 23183231
- [Derived] Gjika E, Beaulieu JY, Vakalopoulos K, Gauthier M, Bouvet C, Gonzalez A, Morello V, Steiger C, Hirsiger S, Lipsky BA, Uckay I. Two weeks versus four weeks of antibiotic therapy after surgical drainage for native joint bacterial arthritis: a prospective, randomised, non-inferiority trial. Ann Rheum Dis. 2019 Aug;78(8):1114-1121. doi: 10.1136/annrheumdis-2019-215116. Epub 2019 Apr 16. PMID 30992295